CLINICAL TRIAL: NCT02243111
Title: Evaluation of Lung Doppler Signals (LDS) in Detecting Pulmonary Arterial Hypertension (PAH) in Patients With Systemic Sclerosis (SSc)
Brief Title: Detecting Pulmonary Arterial Hypertension (PAH) in Patients With Systemic Sclerosis (SSc) by Ultrasound
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Echosense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: DOP22_1
Record Dates: First submitted 2014-09-08; First posted 2014-09-17 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2014-06

CONDITIONS: Systemic Sclerosis; Pulmonary Hypertension
Keywords: Systemic sclerosis, pulmonary hypertension
MeSH Terms: conditions — Scleroderma, Systemic; Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doppler ultrasound (Experimental): Recording Doppler signals from the lungs
  Interventions: Radiation: Doppler ultrasound

INTERVENTIONS:
Radiation: Doppler ultrasound — Detecting Doppler signals from the lungs on the right chest wall

SUMMARY:
Doppler signals can be recorded from the lung parenchyma by means of a pulsed Doppler ultrasound system incorporating a special signal processing package; i.e. the transthoracic parametric Doppler (TPD) (EchoSense Ltd., Haifa, Israel). Systemic sclerosis patients often develop pulmonary vascular disease leading to pulmonary hypertension. The TPD system may provide important insight into pulmonary blood vessels characteristics by the LDS signals that are related to pulmonary hypertension.

The TPD performance in detecting PAH in SSc patients will be assessed in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give signed informed consent prior to enrollment
2. Male or female, ≥ 18 years of age
3. Diagnosis of SSc according to 2013 ACR/EULAR SSc Classification Criteria (van den Hoogen 2013): Score ≥ 9.
4. Patients with RHC data available from measurement within 3 weeks prior to TPD assessment
5. No change in or initiation of PAH specific therapy between the last RHC and TPD

Exclusion Criteria:

1. People unable or unwilling to give informed consent.
2. PCWP or LVEDP > 15 mmHg
3. Any PH etiology outside Group 1 (Dana Point, 2008)
4. Pregnant women
5. Patients having severe chest wall deformity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of SSc patients correctly identified with pulmonary hypertension severity in each of the 4 defined groups by RHC. | 12 month
  Analyze Doppler data of 4 SSc groups(according to pulmonary hypertension sevirity ) resulting in typical features. The features will be implemented in a pre-determined diagnostic algorithm that will determine the overall statistical analysis success of the method in comparison to RHC data.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Molad, Principal Investigator — Reumatology department, Rabin medical center
Locations (1):
- Reumatology department, Rabin medical center, Petah Tikva, Israel